CLINICAL TRIAL: NCT00827164
Title: Resistance Training During Radiation Therapy for Pharyngeal or Laryngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ROG-SCCI 09-001-1; UAB IRB X121218021 (Other Grant/Funding Number: American Institute for Cancer Research)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Head and Neck Cancer; Pharyngeal Cancer; Laryngeal Cancer
Keywords: head and neck cancer; resistance training; nutrition counseling; radiation therapy; pharyngeal or laryngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Nutritional Status; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance Training (Experimental): Patient will meet with an exercise specialist once per week for the first 6 weeks. Patients will receive guidance in a safe and appropriate exercise regimen based on specific medical history and preference. An exercise specialist will telephone weekly for consultation and support once per week for the final 6 weeks.
  Interventions: Behavioral: Resistance Training
- Nutrition Counseling (Other): Patients will meet once per week with dietitian for the first 6 weeks in 60 minute sessions. Dietitian will telephone each patient weekly for the final 6 weeks of counseling and support.
  Interventions: Behavioral: Nutrition Counseling

INTERVENTIONS:
Behavioral: Nutrition Counseling — Patients will meet once per week with dietitian for the first 6 weeks in 60 minute sessions. Dietitian will telephone each patient weekly for the final 6 weeks of counseling and support.
  Other Names: nutrition
  Arms: Nutrition Counseling
Behavioral: Resistance Training — Patient will meet with an exercise specialist once per week for the first 6 weeks. Patients will receive guidance in a safe and appropriate exercise regimen based on specific medical history and preference. An exercise specialist will telephone weekly for consultation and support once per week for the final 6 weeks.
  Arms: Resistance Training

SUMMARY:
The purpose of this feasibility study is to examine the effect of resistance training on muscle strength, lean body mass, physical functioning, fatigue, and quality of life in head and neck cancer patients receiving radiation therapy.

DETAILED DESCRIPTION:
Head and neck cancer (HNCa) patients often lose significant body weight and lean mass which is associated with higher mortality, greater fatigue, poorer quality of life, and reduced physical functioning. Because nutritional supplementation may not consistently improve lean body mass, resistance training may be beneficial. HNCa patients experience unique side effects that impact nutritional status, limiting generalization of exercise intervention study results in other cancer types to HNCa patients. Therefore, 44 HNCa patients will be enrolled in a randomized controlled trial with the following study aims:

Primary study aim: Because this pilot proposal is among the first to attempt a randomized controlled exercise trial in HNCa patients, the primary study aim examines feasibility (e.g., study acceptance, recruitment, intervention process evaluation, adherence, adverse events, retention). The investigators hypothesize that study procedures will require minor alterations in future studies.

Secondary study aim #1: Because effect sizes are necessary for planning efficacy trials, the proposal will compare the effect of a 12-week resistance training plus nutritional counseling intervention versus nutritional counseling alone on muscle strength, lean body mass, physical functioning, fatigue, and quality of life in HNCa patients receiving radiation with or without chemotherapy. The investigators hypothesize that patients receiving resistance training with nutritional counseling will demonstrate greater improvements in the outcomes when compared with participants receiving nutritional counseling alone.

Secondary study aim #2: To enhance adherence in future intervention trials, this proposal will determine resistance training and nutritional adherence rates and associated factors among HNCa patients using attendance records, exercise logs, diet records, self-administered survey, and medical record review. The investigators hypothesize that adherence rates will be lower than that of other cancer populations with correlates including demographic, medical, and psychosocial factors.

Assessments will occur at baseline (first week of radiation), week 6 (mid-intervention), and week 12 (post-intervention). Qualitative and quantitative (e.g., rates, 95% confidence intervals) will assess feasibility and mixed model ANOVA will examine group differences. This information is critical for the design of future resistance training efficacy trials in HNCa patients to prevent lean body mass loss in HNCa patients, potentially reducing mortality, minimizing fatigue, and improving physical functioning and quality of life.

ELIGIBILITY:
Inclusion criteria:

* 1st time diagnosis of head and neck cancer (stage I, II, III, or IV; pharyngeal, laryngeal, nasopharyngeal, oral, floor of mouth, tongue, palate, maxillary, or mandibular)
* age 19 to 90 years old
* English speaking
* radiation therapy planned or underway < 1 week
* Karnofsky performance status ≥ 60%, and
* able to stand

Exclusion Criteria:

* dementia or organic brain syndrome
* severe emotional distress
* active schizophrenia
* quadriplegia or loss of use of limbs or torso
* tendon rupture
* muscle tear
* another diagnoses of cancer in the past 5 years, and
* oncologist refuses to allow screening for possible study participation

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of head and neck cancer patients recruited to participate | up to 24 months
  to test the feasibility of a randomized controlled exercise trial in head and neck cancer patients receiving radiation therapy

SECONDARY OUTCOMES:
change in muscle strength | baseline, week 6, and week 12
  dynamometer measurement
Number of patients who adhere to cohort activity schedule | baseline, week 6, and week 12
  completion of exercise or diet recommendations
change in lean body mass | baseline, week 6, week 12
  bioelectrical impedence
change in physical functioning | baseline, week 6, week 12
  physical performance by doing a semi-tandem, tandem, or side by side stance with the feet, an 8 foot walk time, and 5 chair rise and sits
change in fatigue level | baseline, week 6, week 12
  13-item Functional Assessment of Cancer Therapy-Fatigue scale
change in quality of life | baseline, week 6, week 12
  37-item Functional Assessment of Cancer Therapy-Head and Neck scale

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q Rogers, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Rogers LQ, Rao K, Malone J, Kandula P, Ronen O, Markwell SJ, Courneya KS, Robbins KT. Factors associated with quality of life in outpatients with head and neck cancer 6 months after diagnosis. Head Neck. 2009 Sep;31(9):1207-14. doi: 10.1002/hed.21084. PMID 19360748
- [Background] Rogers LQ, Malone J, Rao K, Courneya KS, Fogleman A, Tippey A, Markwell SJ, Robbins KT. Exercise preferences among patients with head and neck cancer: prevalence and associations with quality of life, symptom severity, depression, and rural residence. Head Neck. 2009 Aug;31(8):994-1005. doi: 10.1002/hed.21053. PMID 19340875